CLINICAL TRIAL: NCT05068726
Title: Clinical Utility of Fluoroestradiol F18 PET/CT in Metastatic Breast Cancer Patients With ER-Positive and HER2-Negative Primary Lesions After Progression on First Line Hormonal Therapy
Brief Title: Clinical Utility of FES F18 PET/CT in Metastatic Breast Cancer Patients
Status: Terminated | Type: Observational
Why Stopped: Sponsor discretion (low recruitment rate)
Sponsor: GE Healthcare (Industry)
Collaborators: Simbec-Orion Group (Industry); Medpace, Inc. (Industry); Zionexa (Industry)
Responsible Party: Sponsor
Other Study IDs: GE-280-401
Record Dates: First submitted 2021-09-24; First posted 2021-10-06 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; PET/CT; Cerianna; FES; Fluoroestradiol F-18
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: 18F Fluoroestradiol Radiopharmaceutical with PET/CT — Administration of one dose of 18F FES for PET/CT imaging
  Other Names: Cerianna

SUMMARY:
This is a phase 4, multi-center, open-label, prospective cohort study to evaluate the clinical utility of Fluoroestradiol F18 (Cerianna) PET/CT to guide therapeutic management in ER-positive, HER2-negative metastatic breast cancer patients with progressive disease on first-line standard-of-care hormonal therapy. All patients will undergo a Cerianna PET/CT scan. The treating physician will complete a standardized questionnaire to indicate the second-line therapeutic management plan before the scheduled Cerianna PET/CT. After interpretation of Cerianna PET/CT by local radiologist or nuclear medicine physician, the treating physician will fill out a similar questionnaire to specify the final therapeutic decision. The proportion of patients with a change in therapeutic management plan based on Cerianna PET/CT results will be the primary endpoint. During the study follow-up period of 18 months, data on standard-of-care imaging, treatments/procedures received, and clinical outcomes will be collected. Patients will be asked to complete a health-related quality of life questionnaire at their screening, 6-month, and 18-month visit. Secondary endpoints include visual and quantitative heterogeneity assessment of tumor Cerianna uptake, and PFS rates at 6 months and 18 months after Cerianna PET/CT, which will be assessed between patients with and without a change in therapeutic management plan. Maximum duration of follow-up for each patient: 20 months. First patient first visit to last patient last visit: estimated 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must sign informed consent prior to enrollment in this trial
* The patient is a female ≥18 years old
* Post-menopausal or pre-menopausal patient with known primary breast tumor(s) expressing ER in ≥1% of tumor cells by IHC
* HER2-negative (0, 1+, 2+ fluorescence in situ hybridization (FISH) negative) primary lesion
* MBC with at least 1 identifiable lesion on standard-of-care imaging assessment, outside of the liver, as confirmed by the investigator site
* Patient with progressive disease on 1st line hormonal therapy (Aromatase Inhibitor) with or without a CDK4/6 inhibitor or mechanistic target of rapamycin (mTOR) inhibitor or phosphoinositide 3-kinases (PI3K) inhibitor
* Patient must score at least 0, 1 or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Status
* Life expectancy of at least 12 months
* The patient is planned to undergo a standard-of-care imaging scan (according to National Comprehensive Cancer Network guidelines, e.g., CT and/or bone scan, or fluorodeoxyglucose [FDG]-PET/CT) covering chest, abdomen, and pelvis after date of consent and before Cerianna PET/CT (Visit 2), or the patient has undergone recent standard-of-care imaging before date of consent and is planned to undergo Cerianna PET/CT (Visit 2) no more than 45 days from the standard-of-care imaging scan

Exclusion Criteria:

* Isolated hepatic metastases (taking into account the physiological hepatic high uptake of Cerianna)
* Patient is on tamoxifen/toremifene treatment without 8-week washout, or on fulvestrant treatment without 28-week washout, (may block ER) before Cerianna PET/CT
* Other evolutive malignant disease (non-melanoma skin cancer is allowed) or acute or chronic infectious disease (well-controlled infectious disease is allowed);
* Patient has a history of administered chemotherapy for metastatic disease; prior chemotherapy in the (neo)adjuvant setting is allowed
* Patient with a known allergy to any of the components of Cerianna
* Woman of childbearing age who is not using effective contraception
* Pregnant woman (per the Product Label and ensured using clinic's standard-of-care), or parturient or nursing mother
* Patient presents with any other clinically active, serious, life-threatening disease, medical, or psychiatric condition, and/or who has a life expectancy of <12 months, or for whom study participation may compromise their management; and/or a patient who the investigator judges to be unsuitable for participation in the study for any reason
* Inability to comply with any requirements of the protocol

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Metastatic Breast Cancer Patients with ER-Positive and HER2-Negative Primary Lesions after Progression on First Line Hormonal Therapy
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluate change in therapeutic management plan assessed by comparing pre/post-Cerianna PET/CT treatment selection (based on comparison of the initial management plan and post-Cerianna PET/CT management plan evaluated within 3 weeks). | [Time Frame: Baseline and within 3 weeks after Cerianna PET/CT
  The percentage of subjects with changes in the therapeutic management plan after Cerianna PET/CT with 95% confidence interval will be estimated by comparison of the initial management plan vs. the post-Cerianna PET/CT management plan evaluated within 3 weeks after Cerianna PET/CT.

SECONDARY OUTCOMES:
Number and percentage of lesions detected with Cerianna PET/CT (focal Cerianna uptake, outside the liver, visible above background) in individual patients. | Time Frame: Baseline, Cerianna PET/CT
  Cerianna-uptake score per patient, defined as total number of Cerianna-positive lesions divided by all lesions visible on standard-of-care imaging (e.g., CT and/or bone scan, or FDG-PET/CT) and Cerianna PET/CT (lower scores represent greater ER heterogeneity/ER loss; 0 = a negative scan)
SUV | Time Frame: Baseline, Cerianna PET/CT
  Standard uptake values (SUVs, incl. SUVmax, SUVmean, SUVpeak) of each measurable lesion on Cerianna PET/CT and the inter-lesion variability of Cerianna uptake in individual patients
Heterogeneity | Time Frame: baseline Cerianna PET/CT and within 3 weeks after Cerianna PET/CT
  Association between Cerianna heterogeneity scores (inter-lesion SUV variability and Cerianna-uptake score) and patients with/without change in therapeutic management plan
Confidence | Time Frame: baseline and within 3 weeks after Cerianna PET/CT
  Treating physician's confidence level in the therapeutic management plan (measured on a 10-point scale) and the percent change in confidence level before and after Cerianna PET/CT
Change in management | Timeframe: baseline, 6 months and 18 months after Cerianna PET/CT
  Proportion of patients with a change in actual therapeutic management assessed by comparing the therapeutic management plans to the actual therapeutic management at 6 months and 18 months after Cerianna PET/CT
PFS | Timeframe: baseline, 6 months and 18 months after Cerianna PET/CT
  PFS rate at 6 and 18 months based on heterogeneity in tumor Cerianna uptake. Comparison will be made between patients with and without a change in therapeutic management plan

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie van de Ven, Study Director — GE Healthcare
Locations (24):
- United States (24):
  - Northern Arizona Healthcare, Flagstaff, Arizona
  - TOI Clinical Research, Cerritos, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of Southern California, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - PET/CT Imaging of San Jose, San Jose, California
  - Providence Saint John's Health Center, Santa Monica, California
  - Valley Breast Care, Van Nuys, California
  - Tampa General Hospital Cancer Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - MD Clinics, Shreveport, Louisiana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The New York Presbyterian Hospital-Columbia University Medical Center, New York, New York
  - WakeMed, Cary, North Carolina
  - Duke University, Durham, North Carolina
  - Kettering Health Cancer Center, Kettering, Ohio
  - St. Luke's University Health Network, Allentown, Pennsylvania
  - University of Pennsylvania / Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Baylor Research Institute d/b/a Baylor Scott & White Research Institute, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington